CLINICAL TRIAL: NCT02837263
Title: Pembrolizumab in Combination With Stereotactic Body Radiotherapy for Liver Metastatic Colorectal Cancer
Brief Title: PI Pembro in Combination With Stereotactic Body Radiotherapy for Liver Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UW15063; NCI-2016-01077 (Registry Identifier: NCI Trial ID); 2016-0303 (Other: Institutional Review Board); A534260 (Other: UW Madison); SMPH\MEDICINE\HEM-ONC (Other: UW Madison); Protocol Version 7/12/2018 (Other: UW Madison)
Record Dates: First submitted 2016-07-15; First posted 2016-07-19 (Estimated); Last update posted 2023-06-12 (Actual); Status verified 2023-01

CONDITIONS: Colorectal Cancer; Colorectal Adenocarcinoma; Stage IVA Colorectal Cancer; Stage IVB Colorectal Cancer; Metastatic Carcinoma in the Liver
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Radiosurgery; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SBRT + Pembrolizumab (Experimental): Subjects will receive stereotactic body radiotherapy (SBRT) within 4 weeks of enrollment. Following SBRT, subjects will receive one cycle of pre-operative pembrolizumab given as an IV over approximately 30 minutes. Surgical management to remove all known sites of metastatic disease should occur 2 weeks post pembrolizumab treatment. Approximately 4-8 weeks after surgery subjects will being the second phase of pembrolizumab treatment. They will receive this treatment every 3 weeks (cycle) for 8 more cycles after surgery. Prior to the 5th cycle of pembrolizumab subjects will also have tumor imaging (CT or MRI).
  Interventions: Radiation: Stereotactic body radiotherapy (SBRT); Drug: Pembrolizumab

INTERVENTIONS:
Radiation: Stereotactic body radiotherapy (SBRT) — SBRT treatment will consist of 40-60 Gy delivered in five fractions prescribed to the planning target volume (PVT). Image guidance with MRI, megavoltage CT or cone beam CT scans would be required.
  SBRT will be initiated on Day 0. This should be initiated within 4 weeks of signing informed consent. An additional 2 weeks will be allowed if necessary due to SBRT treatment planning.
  Other Names: Stereotactic Body Radiation Therapy
Drug: Pembrolizumab — Pembrolizumab is a potent and highly selective humanized monoclonal antibody (mAb) of the IgG4/kappa isotype designed to directly block the interaction between PD-1 and its ligands, PD-L1 and PD-L2. KeytrudaTM (pembrolizumab) has recently been approved in the United Stated for the treatment of patients with unresectable or metastatic melanoma and disease progression following ipilumumab and, if BRAF V600 mutation positive, a BRAF inhibitor.
  Other Names: Pembro; Keytruda

SUMMARY:
The purpose of this research study is:

* To find out how safe the study drug, pembrolizumab, is when combined with stereotactic body radiotherapy (SBRT) to the liver.
* To see how well subjects can tolerate treatment with pembrolizumab and SBRT.
* To find out how often colorectal cancer comes back 1 year after surgically removing all known disease and being treated with SBRT and pembrolizumab.

DETAILED DESCRIPTION:
This is a phase 1b feasibility study to evaluate the use of PD-1 blockade in combination with ablative radiotherapy for the treatment of metastatic colorectal cancer (CRC). This study will examine the sequential combination of stereotactic body radiotherapy (SBRT) and pembrolizumab for patients for whom the goal is eradicating all known sites of disease. It is very likely that for many patients the SBRT therapy will be completed following other modalities including operative resection or ablation.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent/assent for the trial
* Be >/= 18 years of age on day of signing consent.
* Have a diagnosis of histologically confirmed metastatic colorectal cancer to the liver (no other sites of metastatic disease)

  * Histologic confirmation of a colorectal primary tumor is acceptable if accompanied by radiographic evidence of metastatic disease
* Tumor must be mismatch repair (MMR) proficient as determined by microsatellite instability or immunohistochemistry for for MMR proteins

  * Microsatellite instability testing must be MSI-stable or MSI-low
  * Or IHC for MMR proteins must demonstrate intact MMR proteins
* Participant must be candidate for SBRT to at least one intrahepatic lesion. There is no limit on the number of intrahepatic lesions the patient may have
* Participant must be a surgical candidate with therapeutic goal of eradicating all known disease with one additional surgery. Portal venous embolization is permitted to ensure resectability.
* Prior resection of extra-hepatic metastatic disease allowed if completed more than 12 months previous to study enrollment and now new extra-hepatic disease has been found
* Have measurable disease based on RECIST 1.1
* Fresh or archived colorectal cancer tissue, preferably from a hepatic metastatic site. Archival tissue is acceptable for enrolled into this study. Participants who have no archival tissue available do not need to undergo a new biopsy solely for the purpose of this study
* Participants must have received at least one prior line or chemotherapy including an irinotecan or oxaliplatin-fluoropyrimidine-based systemic treatment for colorectal cancer
* Have performance status of 0 or 1 on the ECOG Performance Scale
* Demonstrate an adequate organ function as defined in Table 1. These labs should be repeated if not completed within 10 days of SBRT treatment initiation
* Female participants of childbearing potential should have a negative urine or serum pregnancy test within 10 days of initiating SBRT. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Female participants of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication (Reference Section 5.7.2). Participants of childbearing potential are those who have not been surgically sterilized or have not been free from menses for >1 year
* Male participant should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy

Exclusion Criteria:

* Current participation and receiving study therapy or previous participation in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the initiation of SBRT
* Prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 (first day of SBRT treatment) or who has not recovered (i.e. < Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier
* Prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e. < Grade 1 or at baseline) from adverse events due to a previously administered agent. Prior radiotherapy to the liver is not allowed

  * Participants with < Grade 2 neuropathy are an exception to this criterion and may qualify for the study
  * If the participant received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy
* Participant has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the initiation of SBRT
* Participant has a known history of active TB (Bacillus Tuberculosis)
* Hypersensitivity to pembrolizumab or any of its excipients
* Participant has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 (first day or SBRT treatment) or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier
* Participant has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent. Prior radiotherapy to the liver is not allowed. (Notes: Participants with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study. If participant received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.)
* Participant has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
* Participant has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Participants with previously resected brain metastases may participate provided it has been at least 6 months and no CNS progression has been identified.
* Participant has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Participant has known history of, or any evidence of active, non-infectious pneumonitis.
* Participant has an active infection requiring systemic therapy.
* Participant has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the participant's participation for the full duration of the trial, or is not in the best interest of the participant to participate, in the opinion of the treating investigator.
* Participant has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Participant is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Participant has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
* Participant has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Participant has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative or quantitative] is detected).
* Participant has received a live vaccine within 30 days of planned start of study therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-08-11 (Actual); Primary Completion 2021-11-02 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Recurrence rate at 1 year | 1 year
  Determine the recurrence rate at 1 year following clearance of metastatic disease in the setting of treatment with SBRT and pembrolizumab

SECONDARY OUTCOMES:
Time to recurrence estimated using the Kaplan-Meier method | up to 6 years
  The 95% confidence of the median time to recurrence will be calculated using the Brookmeyer-Crowley method
Disease-free survival estimated using the Kaplan-Meier method | up to 6 years
  The 95% confidence of the median time to disease free survival calculated using the Brookmeyer-Crowley method.
Overall survival estimated using the Kaplan-Meier method | up to 6 years
  The 95% confidence of the median time to overall survival calculated using the Brookmeyer-Crowley method.

OTHER OUTCOMES:
PET/MR imaging parameters | 1 year
  Imaging biomarkers (SUVtot, SUVmean, SUVmax) will be summarized using standard descriptive statistics in terms of means, standard deviations, medians, and ranges. Percentage changes in imaging biomarkers will be calculated between assessment time points. Logistic regression analysis will be conducted to evaluate whether changes in imaging biomarkers predict the recurrence rate at 1 year following clearance of metastatic disease.
Tumor-infiltrating lymphocytes | 1 year
  The number of tumor-infiltrating lymphocytes will be summarized in terms of means and standard deviations for each assessment time point. A negative binomial regression or overdispersed Poisson regression model with patient specific random effects will be used to evaluate changes in the number of tumor-infiltrating lymphocytes.
Expression levels of PDL1 | 1 year
  Linear regression analysis will be conducted to examine the correlation between expression levels of PDL1 in colorectal cancer (CRC) liver metastases.

CONTACTS AND LOCATIONS:
Overall Officials: Dustin Deming, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Carbone Cancer Center, Madison, Wisconsin, United States

REFERENCES:
- See also: UW Carbone Cancer Center Home Page — https://cancer.wisc.edu/